CLINICAL TRIAL: NCT04300439
Title: Medico-economic Interest of Single-use Ancillary Efficiency® in Fitting a GMK® Total Knee Arthroplasty (TKA)
Acronym: IMEDUU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: Medacta USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RC18_0423
Record Dates: First submitted 2020-01-16; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Knee Arthropathy
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: metallic reusable ancillary. (Active Comparator): This control group will be constituted of patients who will have the GMK® prosthesis with metallic reusable ancillary.
  Interventions: Device: knee total arthroplasty with two types of ancillaries
- Arm B: Efficiency single use ancillary. (Experimental): This group will be constituted of patients who will have the GMK® prosthesis with Efficiency single use ancillary.
  Interventions: Device: knee total arthroplasty with two types of ancillaries

INTERVENTIONS:
Device: knee total arthroplasty with two types of ancillaries — -For the Arm A, the surgical procedure of knee total arthroplasty will be done with metallic reusable ancillary.
  For the Arm B, the surgical procedure of knee total arthroplasty will be done with Efficiency single use ancillary.

SUMMARY:
Clinical studies on single-use ancillaries are still few; medico-economic benefits have to be assessed regarding their design and use.

A foreseeable increase in the number of surgeries in the future, tends to change the techniques and consequently to question the medico-economic context. Single-use ancillaries attempt to provide solutions to today's imperatives and could be relevant from a global medico-economic point of view.

For the moment, the conventional ancillaries for TKA are reused after sterilization.

The objective of the study is to improve the fluidity of the intervention process with cost control.

DETAILED DESCRIPTION:
After validation of the inclusion criteria, the surgeon will perform the randomization (1:1): single-use ancillary group or conventional ancillary group. Only the medical team and the block staff will be informed about the ancillary group, not the patient.

The use of the single-use ancillary does not induce any modification of the surgical technique for fitting a TKA. The surgical approach is unchanged and is specific to the surgeon. The appearance and use of the single-use ancillary are similar to the conventional ancillary except for the materials used for their design. Please note that a preliminary training at the beginning of the study will be carried out with the different investigators so that they can handle the different medical devices.

In total, 48 participants will be randomized. The medico-economics assessments will be performed for 20 patients (10 per group) by micro-costing to evaluate the preoperative, intraoperative and post-operative costs : reconditioning time, sterilization and transport time, preparation time and duration of intervention. The qualitative score of subjective assessment of the operator's perception of the ancillary measured during the intervention. The participants will evaluate their QOL by completing a questionnaire 3 month and 12 month postoperative. The safety parameters will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patient with gonarthrosis or inflammatory arthrosis of the knee leading to surgical indication for total knee arthroplasty
* Informed patient, able to understand the information, not opposing to participate this protocol
* patient affiliate to social security

Exclusion Criteria:

* Extra-joint Deformation needing bone associated gesture
* Preoperative active or suspected infection
* Local evolutive tumoral pathology
* Medical history with bone gesture on concerned knee
* Patient unable or refusing to give his consentement
* Pregnant woman or in age to be pregnant without use any effective contraceptive method
* Patient under maintenance of justice, tutelage or legal guardianship)
* Presence of any family, sociological, political or geographic situation able to interfere with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Mean production cost of the surgical intervention (total knee arthroplasty) each arm, from an hospital perspective, using a micro-costing approach with items reported in a eCRF | Day 0
  Mean production cost of the surgical intervention in each arm is calculated thanks to 2 steps : 1) Quantification of health resources consumed during the surgical intervention (transport, cleaning, reconditionning sterilization of ancillaries, time spent by medical staff, nurses and materials used. (These data will be collected on a paper sheet and reported in a eCRF for 20 patients (10 per group)) ; 2) Valuation of health resources consumed with hospital cost accounting, mean wages, and purchase prices of materials.

SECONDARY OUTCOMES:
Incremental cost-utility ratio comparing single use ancillary versus reusable ancillary | 1 year
  Incremental cost-utility ratio comparing single use versus reused ancillaries
clinical functional result in each group (Total KSS score) | 1 year postoperative
  Total KSS score
clinical functional result in each arm | 3 months postoperative
  Total KSS score
HKA angle | 1 year postoperative
  HKA angle will be measured using a whole-leg radiograph (X-rays)
HKA angle | 3 months postoperative
  HKA angle will be measured using a whole-leg radiograph (X-rays)
Number of Adverse events in each arm | 1 year postoperative
  All complications related to the material or occurring in the postoperative year will be reported and compared (anemia, phlebitis, hematoma, scar disunity, scar necrosis, nosocomial infection, fracture)
Euroqol EQ-5D-5L quality-of-life questionnaire (5 questions with 5 possible answers) | 1 year postoperative
  Answers to EQ-5D-5L are used to calculate QALYs which represent a measure of survival weighted by health-related quality-of-life factors so that a weight of 0 represents death and a weight of 1 represents the best imaginable health status.
Euroqol EQ-5D-5L quality-of-life questionnaire (5 questions with 5 possible answers) | 3 months postoperative
  Answers to EQ-5D-5L are used to calculate QALYs which represent a measure of survival weighted by health-related quality-of-life factors so that a weight of 0 represents death and a weight of 1 represents the best imaginable health status.
qualitative score of surgeon's perception about ancillary (1-Excellent, 2-Good, 3- Difficult, 4- Unsure) | Day 0
  This qualitative score will be measured during the intervention and will include 4 levels evaluating grip and comfort
  1. Excellent (good position in a few seconds, no doubt)
  2. Good (easy to use for the first time)
  3. Difficult (several attempts, difficult handling, uncomfortable)
  4. Unsure (persistence of doubt during use)
weight of waste | Day 0
  contaminated and uncontaminated waste will be weighed at the exit of the operating room

CONTACTS AND LOCATIONS:
Overall Officials: Mike Persigant, MD, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes (University Hospital of Nantes), Nantes, France

IPD SHARING:
Plan to Share IPD: No